CLINICAL TRIAL: NCT06970067
Title: Co-Creating and Implementing Contextually Responsive Physical Activity Interventions With Middle School Adolescents
Brief Title: Co-Creating Active Middle School Communities to Increase Student Physical Activity
Acronym: AMSC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Deanna Hoelscher (Other)
Collaborators: University of Texas at Austin (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor-Investigator, Deanna Hoelscher, Regional Dean, Professor, The University of Texas Health Science Center, Houston
Organization: The University of Texas Health Science Center, Houston (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-23-1139; 1R01MD019423 (NIH)
Record Dates: First submitted 2025-03-11; First posted 2025-05-14 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Physical Activity
Keywords: physical activity; adolescent health; active transport; active leisure; middle school
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The intervention will be conducted in three middle school catchment areas, with three additional middle school catchment areas with usual programs used as comparison.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical activity intervention co-produced by the community and investigators (Experimental): This intervention will engage multi-sectoral and multi-generational community members and middle school students for co-producing (co-design, co-implementation, and co-evaluation) contextually-responsive intervention strategies to improve access to active transport and leisure in three middle school communities.
  Interventions: Behavioral: Active Middle School Communities
- Usual environmental and programmatic programs (No Intervention): During the trial, three comparison school communities will not receive the intervention and will engage in usual environmental and programmatic programs. After the trial is completed, these schools will receive a modified version of the programs and strategies developed in the intervention arm (delayed intervention).

INTERVENTIONS:
Behavioral: Active Middle School Communities — This intervention will engage multi-sectoral and multi-generational community members and middle school students to co-produce (co-design, co-implementation, and co-evaluation) contextually-responsive intervention strategies to improve access to active transport and leisure, resulting in increased physical activity and decreased risk for chronic disease in middle school communities. This intervention will use community-based participatory methods, with resources provided for changes in the built environment around the school catchment area.
  Arms: Physical activity intervention co-produced by the community and investigators

SUMMARY:
The purpose of this study is to identify community-level barriers and facilitators for active transport and leisure physical activity and to co-create and test the effectiveness and longer-term sustainability of community-based physical activity intervention strategies in middle schools. Participation in this study may help the investigators and scientific community better understand and address child physical activity and health. This study will collect information about middle school children's physical activity behaviors, habits, knowledge, and activity. The UTHealth School of Public Health is leading the study together with the University of Texas at Austin.

DETAILED DESCRIPTION:
Early adolescence is a critical window of opportunity for establishing lifelong physically active lifestyles. During this stage, youth seek autonomy and experience independent mobility. However, steep declines in physical activity occur in adolescence, a trend that continues into adulthood. This is partly due to reduced opportunities for structured exercise and sports in later life relative to childhood. Despite this, most school-based interventions heavily focus on physical education, sports participation, and active recess strategies (i.e., leisure), with less emphasis on promoting utilitarian (transport-based) physical activity.

Interventions prioritizing the entire school community (including students, their families, and school neighborhood residents), and focused on increasing active transport and leisure, might have a more significant and sustainable impact over the lifespan. To be effective and contextually responsive, however, intervention development, implementation, and evaluation must be collaboratively conducted with and through local community members.

This project proposes to conduct a comprehensive and community-engaged mixed methods study to design and test strategies for improving community-wide and individual-level physical activity outcomes in middle school neighborhoods. The specific aims of this study are:

Aim 1. To identify community-level barriers and facilitators for physical activity in middle school communities using a comprehensive mixed methods approach (Delphi method with Group Concept Mapping, geospatial analysis, participatory GIS).

Aim 2. To engage multi-sectoral and multi-generational community actors for co-creating contextually-responsive intervention strategies to improve access to active transport and leisure in middle school communities.

Aim 3. To conduct a first-generation, controlled trial testing the effectiveness of the co-created intervention strategies for improving physical activity outcomes in middle school communities.

Hypothesis 3.1. 12-month pre-post change in daily minutes of moderate- to vigorous-intensity physical activity (MVPA) will be higher among middle school students (grades 6-7) in school communities that implement co-created strategies relative to comparison school communities.

Hypothesis 3.2 (exploratory). Community-based physical activity levels will improve at 12 months in intervention school communities, relative to comparison school communities.

Hypothesis 3.3. (exploratory). The intervention will improve community-level outcomes, including enhanced community norms regarding active travel, collective efficacy for physical activity, and perceived neighborhood traffic and crime safety.

If successful, these strategies can be scaled up to help increase physical activity among middle school children and communities in the U.S. Increased physical activity among middle school youth can lead to higher levels of physical activity throughout the lifespan, potentially decreasing or attenuating chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Parent/guardian and child/adolescent dyads
* Child/adolescent must be enrolled in the 6th grade at participating schools at baseline
* Parent/guardian and child/adolescent must reside in the same household
* Parent/guardian and child/adolescent must reside within the school catchment area (school community)
* Parent/guardian must speak English or Spanish
* Child/adolescent must speak English

Exclusion Criteria:

* Child/adolescent has a condition that precludes or decreases participation in physical activity
* Child/adolescent cannot complete a written survey

Ages: 11 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Child/adolescent physical activity | Baseline, 12 months (initial effectiveness), and 24 months (sustainability)
  Measured using Accelerometry to determine minutes of moderate-to-vigorous- physical activity (MVPA)

SECONDARY OUTCOMES:
Percentage of children/adolescents using active transport to/from school | Data will be collected for 4 years in both fall and spring each year (Years 2-5) for 8 data points.
  Measured using Active Commuting to School Tallies to obtain counts of children/adolescents who walk or bike to or from school compared to all children/adolescents

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas Health Science Center at Houston, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No